CLINICAL TRIAL: NCT00496028
Title: A Phase I, Open-label Study to Assess the Safety and Tolerability of AZD0530 in Combination With Carboplatin and/or Paclitaxel Chemotherapy in Patients With Solid Tumours
Brief Title: Phase I Study in Patients With Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Mary Stuart, MD - Medical Science Director EPT1, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D8180C00023; AZD0530 study 23
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Last update posted 2010-09-22 (Estimated); Status verified 2010-09

CONDITIONS: Neoplasms
Keywords: Solid tumors; locally advanced or Metastatic Cancer suitable for treatment with carboplatin and/or paclitaxel
MeSH Terms: conditions — Neoplasms | interventions — saracatinib; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): AZD0530 + Paclitaxel
  Interventions: Drug: AZD0530; Drug: Paclitaxel
- 2 (Experimental): AZD0530 + Carboplatin
  Interventions: Drug: AZD0530; Drug: Carboplatin
- 3 (Experimental): AZD0530 + Carboplatin + Paclitaxel
  Interventions: Drug: AZD0530; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: AZD0530 — oral tablet
Drug: Carboplatin — intravenous infusion
  Arms: 2; 3
Drug: Paclitaxel — intravenous infusion
  Arms: 1; 3

SUMMARY:
This study will comprise 2 parts, a dose escalation phase and a dose expansion phase. The 2 phases are part of a single study and described by this single protocol. Patients entered into the dose escalation phase will not be entered into the expansion phase. All subjects must be suitable for treatment with either carboplatin and/or paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy > 12 weeks
* Women defined as post-menopausal
* Male or female patients with locally advanced or metastatic cancer suitable for treatment with carboplatin and/or paclitaxel

Exclusion Criteria:

* Inadequate bone marrow reserve
* Inadequate live function, renal function or low haemoglobin
* Unresolved toxicity from anti-cancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2007-03; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of AZD0530 in combination with carboplatin and/or paclitaxel regimens with solid tumours by assessment of AEs, physical examination, BP, pulse, ECG, laboratory findings, PFTs and thoracic CT scans. | Assessed at each visit

SECONDARY OUTCOMES:
To determine the Maximum Tolerated Dose of AZD0530 when administered in combination with carboplatin and/or paclitaxel by assessment of safety and tolerability data generated for each treatment arm. | Assessed at each visit
To make a preliminary evaluation of clinical response by assessment of RECIST evaluation, time to progression and serum tumour markers. | Assessment at end of study
To investigate the PK of AZD0530. paclitaxel and carboplatin when co-administered to patients with solid tumours, by assessment of appropriate PK parameters. | Predetermined timepoints after dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Steinar Aamdal, MD, Principal Investigator — Radium Hospital, Norway; Mary Stuart, MD, Study Director — AstraZeneca
Locations (7):
- France (2):
  - Research Site, Paris
  - Research Site, Pierre-Bénite
- Netherlands (2):
  - Research Site, Amsterdam
  - Research Site, Groningen
- Research Site, Oslo, Norway
- United Kingdom (2):
  - Research Site, Glasgow
  - Research Site, Sutton